CLINICAL TRIAL: NCT06388252
Title: Electrochemotherapy Induces Changes in the Tumor Microenvironment of Cutaneous and Subcutaneous Metastases in Patients With Cutaneous Melanoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: Slovenian Research and Innovation Agency (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: ERID-KSOPR-0049/2023; 0120-297/2023/3 (Other: National Medical Ethics Committee of the Republic of Slovenia)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Cutaneous Malignant Melanoma
Keywords: In-transit melanoma metastases; Cutaneous and subcutaneous melanoma metastases; Electrochemotherapy; Bleomycin; Cysplatin
MeSH Terms: conditions — Melanoma, Cutaneous Malignant | interventions — Electrochemotherapy

STUDY DESIGN:
Intervention Model Description: Electrochemotherapy with intratumoural cysplatin is recommended for smaller (less than 3 cm) and fewer tumours (up to 10 lesions), while electrochemotherapy with intravenous bleomycin is preferable for multiple and larger tumours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrochemotherapy with Intratumoral Cysplatin (Active Comparator): ECT will be performed directly after the intratumorally administration of cysplatin (0,5-2 mg/cm3 tumor). CliniporatorTM (IGEA S.P.A., Carpi, Italy) will be used to apply the pulses (8 pulses, 1300 V/cm, 100 μs, 5 kHz). Triggering of the electrical pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart. The type of electrode used will be selected according to the size and location of the tumors.
  Interventions: Procedure: Electrochemotherapy with Intratumoral Cysplatin
- Electrochemotherapy with Intravenous Bleomycin (Active Comparator): ECT will be performed within 8 - 28 minutes after intravenous bolus administration of bleomycin (15.000 IU/m2 BSA). CliniporatorTM (IGEA S.P.A., Carpi, Italy) will be used to apply the pulses (8 pulses, 1300 V/cm, 100 μs, 5 kHz). Triggering of the electrical pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart. The type of electrode used will be selected according to the size and location of the tumors.
  Interventions: Procedure: Electrochemotherapy with Intravenous Bleomycin

INTERVENTIONS:
Procedure: Electrochemotherapy with Intratumoral Cysplatin — ECT will be performed directly after the intratumorally administration of cysplatin (0,5-2 mg/cm3 tumor). CliniporatorTM (IGEA S.P.A., Carpi, Italy) will be used to apply the pulses (8 pulses, 1300 V/cm, 100 μs, 5 kHz). Triggering of the electrical pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart. The type of electrode used will be selected according to the size and location of the tumors.
  Other Names: Electrochemotherapy with Intravenous Bleomycin
  Arms: Electrochemotherapy with Intratumoral Cysplatin
Procedure: Electrochemotherapy with Intravenous Bleomycin — ECT will be performed within 8 - 28 minutes after intravenous bolus administration of bleomycin (15.000 IU/m2 BSA). CliniporatorTM (IGEA S.P.A., Carpi, Italy) will be used to apply the pulses (8 pulses, 1300 V/cm, 100 μs, 5 kHz). Triggering of the electrical pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart. The type of electrode used will be selected according to the size and location of the tumors.
  Arms: Electrochemotherapy with Intravenous Bleomycin

SUMMARY:
In the last 10 years, the treatment of metastatic cutaneous melanoma has changed dramatically. The new systemic treatment with immunotherapy has led to a dramatic improvement in quality of life and overall survival. Systemic treatment means that the patient receives the drug as an infusion into a vein. Unfortunately, we know that immunotherapy is not equally successful in all patients. Recent studies have shown that the success of the treatment is not only influenced by the cellular composition of the metastasis, but also by its surroundings. This is called tumor microenvironment. Depending on the differences in the composition of this microenvironment, some metastases can be described as immunologically hot and others as immunologically cold. Immunologically hot metastases respond better to immunotherapy than immunologically cold metastases.

Studies have shown that with some interventions we can change the tumor microenvironment from being immune-cold to being immune-hot. Electrochemotherapy is one of the interventions that might improve the efficacy of immunotherapy in cutaneous melanoma. Electrochemotherapy is an established method for the local treatment of tumors, in which only a certain tumor is treated with special electrodes, to which a weak electric current is applied. We hypothesize that electrochemotherapy stimulates the body's own immune response and enables more effective treatment. Since immunotherapy also stimulates the body's own immune response to cutaneous melanoma cells, the interaction of the two drugs could be even more successful. Recent research results support this assumption.

The primary objective is to evaluate the changes in the tumor microenvironment of cutaneous and subcutaneous melanoma metastases induced by electrochemotherapy, based on the histologic analysis of treated and untreated metastases before and after treatment. The secondary aim is to determine whether the changes in the tumor microenvironment differ depending on the chemotherapeutic agent used.

The results will help us to better understand the synergistic effects of electrochemotherapy and immunotherapy on cutaneous melanoma metastases. The combination of systemic immunotherapy and electrochemotherapy could become an important treatment method for patients with metastatic melanoma.

DETAILED DESCRIPTION:
The study is prospective. The primary objective is to evaluate the changes in the tumor microenvironment of cutaneous and subcutaneous melanoma metastases induced by electrochemotherapy (ECT), based on the histologic analysis of treated and untreated metastases before and after treatment. The secondary aim is to determine whether the changes in the tumor microenvironment differ depending on the chemotherapeutic agent used.

In the study 10-15 patients will be enrolled and devided in two arms, ECT with bleomycin and ECT with cysplatin.

ECT will be offered to patients with cuteaneous melanoma and at least 5 in-transit or distant cutaneous and/or subcutaneous melanoma metastases regardless of previous treatments. The decision will be made in a multidisciplinary tumor board. The choice of chemotherapeuthic drug will depend on the size andnumber of lesions to be treated. Inclusion in the study has no influence on the decision regarding the timing of treatment with immunotherapy. Treatment with immunotherapy will later be included as a factor in the statistical analysis.

ECT will be performed according to the standard operating procedures for the treatment of cutaneous and subcutaneous tumors with ECT. ECT will be performed within 8 - 28 minutes after intravenous bolus administration of bleomycin (15.000 IU/m2 BSA) or directly after the intratumorally administration of cysplatin (0,5-2 mg/cm3 tumor). CliniporatorTM (IGEA S.P.A., Carpi, Italy) will be used to apply the pulses (8 pulses, 1300 V/cm, 100 μs, 5 kHz). Triggering of the electrical pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart. The type of electrode used will be selected according to the size and location of the tumors.

One cutaneous/subcutaneous metastasis will be excised before ECT. One treated cutaneous/subcutaneous metastasis will be excised 2-4 and 9-13 days after the procedure. An untreated cutaneous/subcutaneous metastasis will be excised on day 9-13. The excisions will be performed under local anesthesia. All patients will be enrolled in the study after the procedures and the study have been explained to them in detail and they have signed an informed consent form. A venous blood sample will be taken at the same time points (before ECT, 2-4 days and 9-13 days after ECT).

Histological examination, assessment of the degree of regression and the presence of tumor infiltrating lymphocytes (TIL) will be performed according to standardized procedures on 2-3 μm thick tissue sections, previously fixed in formalin and embedded in paraffin (FFPE), stained with the hematoxylin-eosin (HE) staining method.

Immunohistochemical characterization of the tumor microenvironment will be performed on 2-4 μm thick tissue sections pre-fixed in formalin and embedded in paraffin. We will use commercially available primary monoclonal antibodies to define the tumor inflammatory infiltrate, stroma and vasculature. We will use the following antibodies: CD3, CD4, CD8, CD56, CD163, FoxP3, ERG, PGM1, CD274 (PD-L1). The choice of antibodies used and the method of pathohistologic analysis may change depending on the results. Specific binding of primary antibodies will be visualized using the recommended three-step detection system OptiView DAB IHC Detection Kit (Cat. No. 760-700; manufactured by Ventana ROCHE inc., Tucson, AZ, USA) according to the manufacturer's instructions. The analysis will be performed by two independent pathologists.

We will also collect the information about previous treatments for cutaneous melanoma and photographic documentation of the effectiveness of ECT treatment. Patients will also fill out internationally recognized, validated quality of life questionnaires (EORTC QLQ-C 30 and EQ-5D-5L) at entollment, after ECT, 3 months, 6 months and 12 months after ECT and then once a year during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* more than 4 cytologically and/or histologically confirmed intransit or distant cutaneous/subcutaneous cutaneous melanoma metastases
* ECT should be proposed as a treatment in the multidisciplinary tumor board
* cutaneous/subcutaneous melanoma metastases, that can be excised under local anesthesia with primary wound closure, minimal morbidity of the procedure (risk of complications < 5%) and nocosmetic or functional consequences of the procedure
* stage IIIB, IIIC or IV of the disease
* age over 18 years
* performance status World Health Organization more than 2
* patients must give informed consent

Exclusion Criteria:

* age less than 18 years
* polimorbidity
* performance status World Health Organization more than 2
* high risk for intervention under general anesthesia;
* wound closure would require coverage with a skin graft or local flap;
* undesirable cosmetic or functional consequences would be expected (face, extensor side of joints)
* patients incapable of understanding the aim of the study or disagree with the entering into the clinical study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the tumor microenvironment of cutaneoys and subcutaneousm melanoma metastases induced by electrochemotherapy | before ECT, 2-4 and 9-13 days after the ECT
  The primary objective is to investigate the changes in the tumor microenvironment of cutaneous and subcutaneous melanoma metastases induced by electrochemotherapy, based on the histological evaluation of treated and untreated metastases before and after treatment.

SECONDARY OUTCOMES:
Diferrent changes in the tumor microenvironment induced by electrochemotherapy with bleomycin or cysplatin | before ECT, 2-4 and 9-13 days after the ECT
  The secondary aim is to determine whether the changes in the tumor microenviroment differ depending on the chemotherapeutic agent used - bleomycin intravenously or cysplatin intratumorally

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Perić, Principal Investigator — Dep. of Surgical Oncology, Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zadnik V, Primic Zakelj M, Lokar K, Jarm K, Ivanus U, Zagar T. Cancer burden in slovenia with the time trends analysis. Radiol Oncol. 2017 Feb 22;51(1):47-55. doi: 10.1515/raon-2017-0008. eCollection 2017 Mar 1. PMID 28265232
- [Background] Littman DR. Releasing the Brakes on Cancer Immunotherapy. Cell. 2015 Sep 10;162(6):1186-90. doi: 10.1016/j.cell.2015.08.038. PMID 26359975
- [Background] Goggins CA, Khachemoune A. The use of electrochemotherapy in combination with immunotherapy in the treatment of metastatic melanoma: a focused review. Int J Dermatol. 2019 Aug;58(8):865-870. doi: 10.1111/ijd.14314. Epub 2018 Nov 26. PMID 30479009
- [Background] Garbe C, Amaral T, Peris K, Hauschild A, Arenberger P, Basset-Seguin N, Bastholt L, Bataille V, Del Marmol V, Dreno B, Fargnoli MC, Forsea AM, Grob JJ, Hoeller C, Kaufmann R, Kelleners-Smeets N, Lallas A, Lebbe C, Lytvynenko B, Malvehy J, Moreno-Ramirez D, Nathan P, Pellacani G, Saiag P, Stratigos AJ, Van Akkooi ACJ, Vieira R, Zalaudek I, Lorigan P; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO), and the European Organization for Research and Treatment of Cancer (EORTC). European consensus-based interdisciplinary guideline for melanoma. Part 2: Treatment - Update 2022. Eur J Cancer. 2022 Jul;170:256-284. doi: 10.1016/j.ejca.2022.04.018. Epub 2022 May 24. PMID 35623961
- [Background] Quaglino P, Mortera C, Osella-Abate S, Barberis M, Illengo M, Rissone M, Savoia P, Bernengo MG. Electrochemotherapy with intravenous bleomycin in the local treatment of skin melanoma metastases. Ann Surg Oncol. 2008 Aug;15(8):2215-22. doi: 10.1245/s10434-008-9976-0. Epub 2008 May 23. PMID 18498012
- [Background] Kunte C, Letule V, Gehl J, Dahlstroem K, Curatolo P, Rotunno R, Muir T, Occhini A, Bertino G, Powell B, Saxinger W, Lechner G, Liew SH, Pritchard-Jones R, Rutkowski P, Zdzienicki M, Mowatt D, Sykes AJ, Orlando A, Mitsala G, Rossi CR, Campana L, Brizio M, de Terlizzi F, Quaglino P, Odili J; InspECT (the International Network for Sharing Practices on Electrochemotherapy). Electrochemotherapy in the treatment of metastatic malignant melanoma: a prospective cohort study by InspECT. Br J Dermatol. 2017 Jun;176(6):1475-1485. doi: 10.1111/bjd.15340. Epub 2017 Apr 26. PMID 28118487
- [Background] Campana LG, Valpione S, Mocellin S, Sundararajan R, Granziera E, Sartore L, Chiarion-Sileni V, Rossi CR. Electrochemotherapy for disseminated superficial metastases from malignant melanoma. Br J Surg. 2012 Jun;99(6):821-30. doi: 10.1002/bjs.8749. Epub 2012 Apr 17. PMID 22508342
- [Background] Cadossi R, Ronchetti M, Cadossi M. Locally enhanced chemotherapy by electroporation: clinical experiences and perspective of use of electrochemotherapy. Future Oncol. 2014 Apr;10(5):877-90. doi: 10.2217/fon.13.235. PMID 24799067
- [Background] Mali B, Jarm T, Snoj M, Sersa G, Miklavcic D. Antitumor effectiveness of electrochemotherapy: a systematic review and meta-analysis. Eur J Surg Oncol. 2013 Jan;39(1):4-16. doi: 10.1016/j.ejso.2012.08.016. Epub 2012 Sep 11. PMID 22980492
- [Background] Gehl J, Sersa G, Matthiessen LW, Muir T, Soden D, Occhini A, Quaglino P, Curatolo P, Campana LG, Kunte C, Clover AJP, Bertino G, Farricha V, Odili J, Dahlstrom K, Benazzo M, Mir LM. Updated standard operating procedures for electrochemotherapy of cutaneous tumours and skin metastases. Acta Oncol. 2018 Jul;57(7):874-882. doi: 10.1080/0284186X.2018.1454602. Epub 2018 Mar 25. PMID 29577784
- [Background] Sersa G, Teissie J, Cemazar M, Signori E, Kamensek U, Marshall G, Miklavcic D. Electrochemotherapy of tumors as in situ vaccination boosted by immunogene electrotransfer. Cancer Immunol Immunother. 2015 Oct;64(10):1315-27. doi: 10.1007/s00262-015-1724-2. Epub 2015 Jun 12. PMID 26067277
- [Background] Polajzer T, Jarm T, Miklavcic D. Analysis of damage-associated molecular pattern molecules due to electroporation of cells in vitro. Radiol Oncol. 2020 Jul 29;54(3):317-328. doi: 10.2478/raon-2020-0047. PMID 32726295
- [Background] Sersa G, Ursic K, Cemazar M, Heller R, Bosnjak M, Campana LG. Biological factors of the tumour response to electrochemotherapy: Review of the evidence and a research roadmap. Eur J Surg Oncol. 2021 Aug;47(8):1836-1846. doi: 10.1016/j.ejso.2021.03.229. Epub 2021 Mar 11. PMID 33726951
- [Background] Ursic K, Kos S, Kamensek U, Cemazar M, Miceska S, Markelc B, Bucek S, Staresinic B, Kloboves Prevodnik V, Heller R, Sersa G. Potentiation of electrochemotherapy effectiveness by immunostimulation with IL-12 gene electrotransfer in mice is dependent on tumor immune status. J Control Release. 2021 Apr 10;332:623-635. doi: 10.1016/j.jconrel.2021.03.009. Epub 2021 Mar 8. PMID 33705828
- [Background] Tremble LF, O'Brien MA, Soden DM, Forde PF. Electrochemotherapy with cisplatin increases survival and induces immunogenic responses in murine models of lung cancer and colorectal cancer. Cancer Lett. 2019 Feb 1;442:475-482. doi: 10.1016/j.canlet.2018.11.015. Epub 2018 Nov 22. PMID 30472183
- [Background] Justesen TF, Orhan A, Raskov H, Nolsoe C, Gogenur I. Electroporation and Immunotherapy-Unleashing the Abscopal Effect. Cancers (Basel). 2022 Jun 10;14(12):2876. doi: 10.3390/cancers14122876. PMID 35740542
- [Background] Falk H, Lambaa S, Johannesen HH, Wooler G, Venzo A, Gehl J. Electrochemotherapy and calcium electroporation inducing a systemic immune response with local and distant remission of tumors in a patient with malignant melanoma - a case report. Acta Oncol. 2017 Aug;56(8):1126-1131. doi: 10.1080/0284186X.2017.1290274. Epub 2017 Feb 22. No abstract available. PMID 28562201
- [Background] Tetzlaff MT, Messina JL, Stein JE, Xu X, Amaria RN, Blank CU, van de Wiel BA, Ferguson PM, Rawson RV, Ross MI, Spillane AJ, Gershenwald JE, Saw RPM, van Akkooi ACJ, van Houdt WJ, Mitchell TC, Menzies AM, Long GV, Wargo JA, Davies MA, Prieto VG, Taube JM, Scolyer RA. Pathological assessment of resection specimens after neoadjuvant therapy for metastatic melanoma. Ann Oncol. 2018 Aug 1;29(8):1861-1868. doi: 10.1093/annonc/mdy226. PMID 29945191
- [Background] Di Gennaro P, Gerlini G, Urso C, Sestini S, Brandani P, Pimpinelli N, Borgognoni L. CD4+FOXP3+ T regulatory cells decrease and CD3+CD8+ T cells recruitment in TILs from melanoma metastases after electrochemotherapy. Clin Exp Metastasis. 2016 Dec;33(8):787-798. doi: 10.1007/s10585-016-9814-x. Epub 2016 Jul 30. PMID 27475809
- [Background] Bigi L, Galdo G, Cesinaro AM, Vaschieri C, Marconi A, Pincelli C, Fantini F. Electrochemotherapy induces apoptotic death in melanoma metastases: a histologic and immunohistochemical investigation. Clin Cosmet Investig Dermatol. 2016 Nov 23;9:451-459. doi: 10.2147/CCID.S115984. eCollection 2016. PMID 27920565
- [Background] Steele MM, Jaiswal A, Delclaux I, Dryg ID, Murugan D, Femel J, Son S, du Bois H, Hill C, Leachman SA, Chang YH, Coussens LM, Anandasabapathy N, Lund AW. T cell egress via lymphatic vessels is tuned by antigen encounter and limits tumor control. Nat Immunol. 2023 Apr;24(4):664-675. doi: 10.1038/s41590-023-01443-y. Epub 2023 Feb 27. PMID 36849745
- [Background] Dimitrakopoulou-Strauss A. Monitoring of patients with metastatic melanoma treated with immune checkpoint inhibitors using PET-CT. Cancer Immunol Immunother. 2019 May;68(5):813-822. doi: 10.1007/s00262-018-2229-6. Epub 2018 Aug 19. PMID 30123922
- [Background] Weiss SA, Wolchok JD, Sznol M. Immunotherapy of Melanoma: Facts and Hopes. Clin Cancer Res. 2019 Sep 1;25(17):5191-5201. doi: 10.1158/1078-0432.CCR-18-1550. Epub 2019 Mar 28. PMID 30923036
- [Background] Campana LG, Peric B, Mascherini M, Spina R, Kunte C, Kis E, Rozsa P, Quaglino P, Jones RP, Clover AJP, Curatolo P, Giorgione R, Cemazar M, Terlizzi F, Bosnjak M, Sersa G. Combination of Pembrolizumab with Electrochemotherapy in Cutaneous Metastases from Melanoma: A Comparative Retrospective Study from the InspECT and Slovenian Cancer Registry. Cancers (Basel). 2021 Aug 25;13(17):4289. doi: 10.3390/cancers13174289. PMID 34503099
- [Background] Heppt MV, Eigentler TK, Kahler KC, Herbst RA, Goppner D, Gambichler T, Ulrich J, Dippel E, Loquai C, Schell B, Schilling B, Schad SG, Schultz ES, Matheis F, Tietze JK, Berking C. Immune checkpoint blockade with concurrent electrochemotherapy in advanced melanoma: a retrospective multicenter analysis. Cancer Immunol Immunother. 2016 Aug;65(8):951-9. doi: 10.1007/s00262-016-1856-z. Epub 2016 Jun 13. PMID 27294607
- [Background] Mozzillo N, Simeone E, Benedetto L, Curvietto M, Giannarelli D, Gentilcore G, Camerlingo R, Capone M, Madonna G, Festino L, Caraco C, Di Monta G, Marone U, Di Marzo M, Grimaldi AM, Mori S, Ciliberto G, Ascierto PA. Assessing a novel immuno-oncology-based combination therapy: Ipilimumab plus electrochemotherapy. Oncoimmunology. 2015 May 22;4(6):e1008842. doi: 10.1080/2162402X.2015.1008842. eCollection 2015 Jun. PMID 26155423

DOCUMENTS (1):
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT06388252/ICF_000.pdf